CLINICAL TRIAL: NCT01106521
Title: A Multicentre Registry Study of Permanent Breast Seed Implant (PBSI) for Early Stage Breast Cancers.
Brief Title: A Registry Study of Permanent Breast Seed Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: West Penn Allegheny Health System (Other); British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Dr. Eric Leung, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBSI Registry
Record Dates: First submitted 2010-04-09; First posted 2010-04-20 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Breast Neoplasms
Keywords: Infiltrating ductal carcinoma; Brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PBSI (Experimental): PBSI is a form of accelerated partial breast irradiation involving the insertion of 103-palladium stranded seeds under ultra-sound guidance and light sedation after CT planning in lieu of whole breast adjuvant radiotherapy.
  Interventions: Radiation: Permanent breast seeds implant

INTERVENTIONS:
Radiation: Permanent breast seeds implant — Patients are pre-planned using CT simulation. Implant is realised under light sedation and local freezing. Stranded seeds are inserted using a brachytherapy template that is immobilised to the planned target volume using a 'localization' needle. Patients is released the same day and Quality Assurance involves a 2 months post-implant CT
  Other Names: Artemend

SUMMARY:
Women found to have early stage breast cancer will have their cancer surgically removed followed by radiation treatment to the entire breast, five times per week for several weeks. The radiation treatment prevents the cancer from growing back but creates skin burns. Several studies have showed that it is nor necessary treating the whole breast.

The investigators team has pioneered a new therapy realizing the permanent implantation of tiny radioactive seeds into the surgical cavity in a single one hour procedure under light anesthesia. Patients live a normal life while receiving the radiation treatment. The results of a first clinical trial on 67 patients shows that the treatment is well tolerate and efficient. The purpose of the study is to offer the treatment in several places and to increase the cohort of patient to 420 to capture rare complications if any.

DETAILED DESCRIPTION:
For early stage breast cancer, accelerated partial breast irradiation is an alternative treatment option to whole breast irradiation after breast conserving surgery. Our group has previously reported results of a Phase I/II study of permanent breast seed implant (PBSI) using palladium-103 seeds as an alternative to whole breast radiotherapy for well selected breast cancer patients. The procedure is realised in a single session under light sedation and local freezing. After a median FU of 54 months no patients has recurred on a cohort of 67 patients, and acute of delayed side effect compared favourably to external beam radiotherapy.

Yet this study was a single centre study and the sample size did not allow evaluating appropriately the risk of serious adverse events (SAE). The current study propose evaluating SAE on a multicentre and larger cohort of 420 patients.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed histological diagnosis of invasive breast carcinoma
* Treated by breast conserving surgery with axillary node dissection (with a minimum of 6 nodes sampled) or sentinel lymph node biopsy
* Surgical margins clear over or equal to 2 mm
* A maximum tumor size of 3 cm
* Age >= 50 years old
* ECOG performance status of 0 or 1
* Informed consent signed

Exclusion Criteria:

* Previous history of cancer other than curable skin SCC or Tis or T1 cervix
* Patient receiving anti-coagulant that cannot be stopped two weeks prior PBSI
* Autoimmune disorder
* Diabetes insulin-dependant
* Pregnancy
* Breast implants
* Psychiatric or addictive disorder that would preclude attending follow-up
* Post-operative breast infection
* Suspicious remaining microcalcification on post-surgery mammogram (unless biopsy proven benign)
* Lobular features on histology (pure or mixed) or sarcoma histology
* Node positive on axillary dissection or in the sentinel lymph node biopsy
* Extensive in situ carcinoma
* Multicentric disease (in more than one quadrant or separated by 2 cm or more)
* Paget's disease of the nipple
* Metastases
* Patients presenting a post-surgical fluid cavity ≥ 2.5 cm in diameter in any dimension as determined on the planning US
* Clear delineation of the target volume on CT is not possible
* Having a volume to be implanted over 120cc
* Having a target volume too close to skin such that the 85% isodose overlaps the skin surface)
* Having a target volume too close to the chest wall, such that there is a risk of perforating the chest wall

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-03; Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | Initial and then yearly up to 5 years
  Serious Adverse Events (SAE) is an unintended sign, symptom, or syndrome illness that occurs during the period of observation in the clinical study and that is life threatening or result in death. SAE will be coded using the NCI CTC V3.0 scale and corresponds to grade 4 or 5 signs or symptoms.

SECONDARY OUTCOMES:
Breast cancer local recurrence | Yearly up to 10 years
  Ipsilateral in-breast or chest wall recurrence is defined as evidence of invasive or in situ breast cancer (except LCIS) in the ipsilateral breast. Patients will have a biopsy of the suspicious lesion to confirm the diagnosis with documentation of the location.
Regional recurrence | Yearly up to 10 years
  Regional recurrence is defined as the development of tumor in regional nodes as well as the soft tissue of the ipsilateral axilla after axillary dissection. The regional recurrence is suspected on imaging and/or clinical symptoms and must be documented with fine needle aspiration. Also the localisation of the nodal recurrence must be reported (internal mammary chain, supra-clavicular area or axilla).
Metastases | Yearly up to 10 years
  Distant recurrence is defined as evidence of tumor in any area of the body. The metastasis recurrence should be proved by appropriate imaging, biopsy or fine needle aspiration
PBSI side effects | After procedure
  Any toxicity related to the radiation treatment, including skin and subcutaneous, or any other organ in case of seed migration will be coded using the NCI common toxicity criteria version 3.0 scale.
PBSI side effects | At 2 months
  Any toxicity related to the radiation treatment, including skin and subcutaneous, or any other organ in case of seed migration will be coded using the NCI common toxicity criteria version 3.0 scale.
PBSI side effect | At 6 months
  Any toxicity related to the radiation treatment, including skin and subcutaneous, or any other organ in case of seed migration will be coded using the NCI common toxicity criteria version 3.0 scale.
PBSI side effect | Yearly up to 10 years
  Any toxicity related to the radiation treatment, including skin and subcutaneous, or any other organ in case of seed migration will be coded using the NCI common toxicity criteria version 3.0 scale. Fat necrosis will be diagnosed either by mammography or clinically (prolonged indurations and pain in the area of seeds implantation without evidence of infection).
Cosmetic outcome | Yearly up to 10 years
  Cosmetic results will be evaluated at each follow-up visit by the treating radiation oncologist. An excellent cosmetic result score is assigned when the treated breast looked essentially the same as the contralateral breast (as it relates to radiation effects). A good cosmetic score is assigned for minimal but identifiable radiation effects of the treated breast. A fair score means significant radiation effects were readily observable. A poor score is used for severe sequelae of breast tissue secondary to radiation effects.
Survival | Yearly up to 10 years
  Patient survival, either free of cancer or with disease present will be recorded at follow-up appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leung, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Keller BM, Pignol JP, Rakovitch E, Sankreacha R, O'Brien P. A radiation badge survey for family members living with patients treated with a (103)Pd permanent breast seed implant. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):267-71. doi: 10.1016/j.ijrobp.2007.08.006. Epub 2007 Oct 29. PMID 17967512
- [Background] Keller B, Sankreacha R, Rakovitch E, O'brien P, Pignol JP. A permanent breast seed implant as partial breast radiation therapy for early-stage patients: a comparison of palladium-103 and iodine-125 isotopes based on radiation safety considerations. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):358-65. doi: 10.1016/j.ijrobp.2004.10.014. PMID 15890575
- [Result] Pignol JP, Rakovitch E, Keller BM, Sankreacha R, Chartier C. Tolerance and acceptance results of a palladium-103 permanent breast seed implant Phase I/II study. Int J Radiat Oncol Biol Phys. 2009 Apr 1;73(5):1482-8. doi: 10.1016/j.ijrobp.2008.06.1945. Epub 2008 Oct 18. PMID 18930602
- [Result] Pignol JP, Keller B, Rakovitch E, Sankreacha R, Easton H, Que W. First report of a permanent breast 103Pd seed implant as adjuvant radiation treatment for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):176-81. doi: 10.1016/j.ijrobp.2005.06.031. Epub 2005 Sep 22. PMID 16182464